CLINICAL TRIAL: NCT01406158
Title: A Phase 1, Open-Label, Randomized, Single Dose, 3-Way Crossover Study to Assess the Relative Bioavailability of Solifenacin Liquid Suspension 10 mg (Formulation B) Versus Solifenacin Liquid Suspension 10 mg (Formulation A) and to Assess the Relative Bioavailability of Solifenacin Liquid Suspension 10 mg (Formulation A and B) Versus the VESIcare (Solifenacin Succinate) 10 mg Tablet in Healthy Volunteers
Brief Title: A Study in Healthy Volunteers Comparing Two Different Liquid Formulations of Solifenacin With Each Other and With the Tablet Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 905-CL-080
Record Dates: First submitted 2011-07-14; First posted 2011-08-01 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Pharmacokinetics of Solifenacin Succinate; Healthy Volunteers
Keywords: Solifenacin succinate; VESIcare; Healthy Volunteers; YM905
MeSH Terms: interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental)
  Interventions: Drug: Solifenacin Succinate Formulation A
- Treatment B (Experimental)
  Interventions: Drug: Solifenacin Succinate Formulation B
- Treatment T (Experimental)
  Interventions: Drug: Solifenacin Succinate

INTERVENTIONS:
Drug: Solifenacin Succinate Formulation A — oral suspension
  Other Names: YM905
  Arms: Treatment A
Drug: Solifenacin Succinate Formulation B — oral suspension
  Other Names: YM905
  Arms: Treatment B
Drug: Solifenacin Succinate — oral tablet
  Other Names: VESIcare; YM905
  Arms: Treatment T

SUMMARY:
A study in healthy volunteers comparing two different liquid formulations of solifenacin with each other and with the tablet formulation.

DETAILED DESCRIPTION:
Subjects will be randomized to one of six treatment sequences. The treatments will be separated by a minimum of 13 days between dosing.

Study drug will be administered after an overnight fast, and food will be restricted for an additional four hours after dosing. Except for the water provided with dosing, water will be restricted only during the hour before and the hour after dosing.

Subjects will stay at the study site for the first three days of each treatment period. Subjects will return to the study center each morning at the same time of the day for Days 4 through 11 of each study period for the pharmacokinetic blood draw and vital signs. Subjects will be in the study for at least 40 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject weighs at least 45 kg, and has a body mass index of 18 to 32 kg/m2
* Subject has a normal 12-lead electrocardiogram (ECG)
* Subject, if female, must be at least 2 years postmenopausal, surgically sterile, or practicing effective birth control, and is not pregnant or lactating
* Subject has good venous access

Exclusion Criteria:

* The subject has a history of any clinically significant disease or malignancy with the exception of non-melanoma skin cancer
* The subject has a history of or currently has evidence of urinary retention, gastric retention, or uncontrolled narrow-angle-glaucoma
* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* The subject has a known hypersensitivity to VESIcare® or any of the excipients in the formulations, or the subject has a history of severe allergic or anaphylactic reactions
* The subject has a history of consuming more than 15 units of alcoholic beverages per week, or has a history of alcoholism or substance abuse within the past two years prior to screening (Note: one unit = 12 ounces of beer, 4 ounces of wine, or 1 ounce of spirits)
* The subject has used tobacco containing products or nicotine containing products within past six months
* The subject has a supine mean systolic blood pressure < 90 or > 160 mmHg and a mean diastolic blood pressure < 50 or > 90 mmHg, or pulse rate < 40 or >100 beats per minute
* The subject is known to be positive for human immunodeficiency virus antibody
* The subject has a positive test for hepatitis C antibody or hepatitis B antigen
* The subject's laboratory test results are outside the normal limits and considered to be clinically significant
* The subject has had treatment with prescription or non-prescription drugs, including complementary and alternative medicines or over-the-counter medications, with the exception of hormonal contraceptives, hormone replacement therapy, and occasional use of acetaminophen within 14 days prior to inclusion into the study
* The subject anticipates an inability to abstain from alcohol or caffeine use throughout the duration of the study or from grapefruit, Seville oranges, star fruit, or any products containing these items from throughout the duration of the study
* The subject has received an experimental agent within past 30 days or ten half-lives, whichever is longer
* The subject has had any significant blood loss
* The subject has any clinically significant history of gastrointestinal symptoms such as nausea, abdominal discomfort or upset, or heartburn in the four weeks prior to clinic admission, or a history of any gastrointestinal surgery except for appendectomy or cholecystectomy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic assessment of AUC and maximum concentration (Cmax) through the analysis of blood samples | Up to Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States